CLINICAL TRIAL: NCT06470204
Title: Infiltration Between the Popliteal Artery and Capsule of the Knee Block With Adductor Canal Block With Ropivacaine vs Ropivacaine and Dexamethasone in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Dexamethasone for iPACK Block With ACB in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7/2024
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine (Active Comparator): iPACK Block + ACB with Ropivacaine
  Interventions: Drug: Ropivacaine
- Ropivacaine + Dexamethasone (Active Comparator): iPACK Block + ACB with Ropivacaine + Dexamethasone
  Interventions: Drug: Ropivacaine+Dexamethasone

INTERVENTIONS:
Drug: Ropivacaine — Ultrasound-guided iPACK block + ACB - 2 x (20ml 0,2% ropivacaine + 2ml 0.9% NaCl)
  Arms: Ropivacaine
Drug: Ropivacaine+Dexamethasone — Ultrasound-guided iPACK block + ACB - 2 x (20ml 0,2% ropivacaine + 2mg Dexamethasone)
  Arms: Ropivacaine + Dexamethasone

SUMMARY:
Effect of adding Dexamethasone to Infiltration between the Popliteal Artery and Capsule of the Knee Block with ACB in Patients undergoing Total Knee Arthroplasty

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most common orthopaedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prostheses. Regional anaesthesia methods may be performed to reduce the inflammatory response, opioid consumption, and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total hip arthroplasty
* patients aged >65 and <100 years
* patients able to provide informed consent
* patients able to reliably report symptoms to the research team

Exclusion Criteria:

* inability to provide first-party consent due to cognitive impairment or a language barrier

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Total Opioid Consumption | 48 hours after surgery
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 4 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 8 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 12 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 48 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Nerve damage [range 0-4] | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
glucose | 12 hours after surgery
  blood glucose level
glucose | 24 hours after surgery
  blood glucose level
glucose | 48 hours after surgery
  blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to eligible researchers following the trial completion
Time Frame: Following the trial completion
Access Criteria: Elligible researcher